CLINICAL TRIAL: NCT05375981
Title: Magnet Ingestion in Children: a Prospective Surveillance Study
Brief Title: MAGNET Ingestion in Children
Acronym: MAGNETIC
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CHI1116
Record Dates: First submitted 2022-05-04; First posted 2022-05-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Foreign Bodies
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One year national observational surveillance study of children who ingest a magnetic foreign body

DETAILED DESCRIPTION:
The study aims to understand the incidence, management and outcomes of children who ingest a magnetic foreign body.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic foreign body ingestion
* 16 years of age or less

Exclusion Criteria:

* Non ingested foreign body

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Definite magnetic foreign body ingestion in children <16yrs
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of MAGNETIC Foreign Body Ingestion | Over 1 year from May 1st 2022

SECONDARY OUTCOMES:
Investigations and management of magnetic foreign body ingestion | Up to 28 days following ingestion
  What investigations and treatments these children had
Outcomes of magnetic foreign body ingestion | Up to 28 days following ingestion
  What the outcomes were

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton Children's Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No